CLINICAL TRIAL: NCT02360475
Title: An Observer-blind Study to Assess the Safety, Reactogenicity and Immunogenicity of Different Formulations of GSK Biologicals' Investigational RSV Vaccine (GSK3003891A), in Healthy Women
Brief Title: Safety, Reactogenicity and Immunogenicity Study of Different Formulations of GlaxoSmithKline (GSK) Biologicals' Investigational RSV Vaccine (GSK3003891A), in Healthy Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201510; 2014-002688-14 (EudraCT Number)
Record Dates: First submitted 2015-01-29; First posted 2015-02-10 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Vaccine; Immunogenicity; Safety; Respiratory syncytial virus (RSV); Reactogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (4):
- RSV vaccine formulation 1 Group (Experimental): Subjects in this group will receive a single dose of formulation 1 of the RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003895A (formulation 1)
- RSV vaccine formulation 2 Group (Experimental): Subjects in this group will receive a single dose of formulation 2 of RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003898A (formulation 2)
- RSV vaccine formulation 3 Group (Experimental): Subjects in this group will receive a single dose of formulation 3 of RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003899A (formulation 3)
- Boostrix Group (Active Comparator): Subjects in this group will receive a single dose of Boostrix
  Interventions: Biological: Boostrix

INTERVENTIONS:
Biological: RSV vaccine GSK3003895A (formulation 1) — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm
  Arms: RSV vaccine formulation 1 Group
Biological: RSV vaccine GSK3003898A (formulation 2) — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm
  Arms: RSV vaccine formulation 2 Group
Biological: RSV vaccine GSK3003899A (formulation 3) — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm
  Arms: RSV vaccine formulation 3 Group
Biological: Boostrix — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm
  Arms: Boostrix Group

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of different formulations of a single intramuscular dose of GSK Biologicals' investigational RSV vaccine, in healthy, non-pregnant women aged 18 to 45 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* Non-pregnant female between, and including, 18 and 45 years of age at the time of study vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * Has practiced adequate contraception for 30 days prior to study vaccination, and
  * Has a negative pregnancy test on the day of study vaccination, and
  * Has agreed to continue adequate contraception during the study period.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days prior to study vaccination, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/ product.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after study vaccination, with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before or after study vaccination.
* Previous experimental vaccination against RSV.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccines.
* History of severe allergic reaction after a previous dose of any tetanus toxoid, diphtheria toxoid, or pertussis antigen-containing vaccine or to any component of Boostrix.
* History of encephalopathy of unknown aetiology occurring within 7 days following a previous vaccination with pertussis-containing vaccine.
* History of any neurological disorders or seizures
* History of transient thrombocytopenia or neurological complications following a previous vaccination against diphtheria and/ or tetanus.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to study vaccination, or planned administration during the study period. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/ or any blood products within the 3 months prior to study vaccination, or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of or current autoimmune disease.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality.
* Malignancy within previous 5 years or lymphoproliferative disorder.
* Current alcohol and/or drug abuse.
* Acute disease and/ or fever at the time of enrolment.
* Hypersensitivity to latex.
* Pregnant or lactating female.
* Planned move to a location that will prohibit participating in the trial until study end.
* Any other condition that the investigator judges may interfere with study procedures or findings.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 507 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2016-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (7):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Austin, Texas
- GSK Investigational Site, Melbourne, Victoria, Australia
- GSK Investigational Site, Hradec Králové, Czechia
- Germany (3):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Dippoldiswalde, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Steff AM, Cadieux-Dion C, de Lannoy G, Prato MK, Czeszak X, Andre B, Ingels DC, Louckx M, Dewe W, Picciolato M, Maleux K, Fissette L, Dieussaert I. Hamster neogenin, a host-cell protein contained in a respiratory syncytial virus candidate vaccine, induces antibody responses in rabbits but not in clinical trial participants. Hum Vaccin Immunother. 2020 Jun 2;16(6):1327-1337. doi: 10.1080/21645515.2019.1693749. Epub 2020 Jan 17. PMID 31951765
- [Derived] Beran J, Lickliter JD, Schwarz TF, Johnson C, Chu L, Domachowske JB, Van Damme P, Withanage K, Fissette LA, David MP, Maleux K, Schmidt AC, Picciolato M, Dieussaert I. Safety and Immunogenicity of 3 Formulations of an Investigational Respiratory Syncytial Virus Vaccine in Nonpregnant Women: Results From 2 Phase 2 Trials. J Infect Dis. 2018 Apr 23;217(10):1616-1625. doi: 10.1093/infdis/jiy065. PMID 29401325
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK3003891A 30 Non-adjuvanted Group: Healthy non-pregnant female subjects between and including 18 and 45 years of age at the time of vaccination received a single dose of the non-adjuvanted 30 µg investigational GSK3003891A vaccine, intramuscularly, in the deltoid region of the non-dominant arm, at Day 0.
- GSK3003891A 60 Non-adjuvanted Group: Healthy non-pregnant female subjects between and including 18 and 45 years of age at the time of vaccination received a single dose of non-adjuvanted 60 µg investigational GSK3003891A vaccine, intramuscularly, in the deltoid region of the non-dominant arm, at Day 0.
- GSK3003891A 60 Adjuvanted Group: Healthy non-pregnant female subjects between and including 18 and 45 years of age at the time of vaccination received a single dose of aluminium-adjuvanted 60 µg investigational GSK3003891A vaccine, intramuscularly, in the deltoid region of the non-dominant arm, at Day 0.
- Boostrix Group: Healthy non-pregnant female subjects between and including 18 and 45 years of age at the time of vaccination received a single dose of Boostrix™ vaccine, intramuscularly, in the deltoid region of the non-dominant arm, at Day 0.
Period: Overall Study
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Started (A total of 507 subjects were screened, but only 500 subjects received vaccination.) | 126 | 124 | 125 | 125
Completed | 122 | 111 | 117 | 120
Not Completed | 4 | 13 | 8 | 5
Not completed — Lost to Follow-up | 4 | 12 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group | Total
Number analyzed (Participants) | 126 | 124 | 125 | 125 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.2 (7.5) | 29.5 (8.2) | 29.1 (7.4) | 29.2 (7.9) | 29.25 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 124 | 125 | 125 | 500
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 5 | 7 | 9 | 9 | 30
  Asian - Central/South Asian Heritage | 0 | 0 | 3 | 0 | 3
  Asian - East Asian Heritage | 1 | 0 | 3 | 0 | 4
  Asian - Japanese Heritage | 1 | 0 | 0 | 0 | 1
  Asian - South East Asian Heritage | 1 | 1 | 6 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  White-Arabic / North African Heritage | 2 | 1 | 2 | 2 | 7
  White-Caucasian/European Heritage | 112 | 114 | 97 | 108 | 431
  Other | 3 | 1 | 5 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = Significant pain at rest, pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling with a maximum diameter greater than 100 millimeters (mm).
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with study vaccines administration documented and with the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 124 | 119 | 124 | 124
Participants
  Any Pain | 62 | 68 | 104 | 104
  Grade 3 Pain | 1 | 2 | 9 | 3
  Any Redness | 6 | 3 | 8 | 6
  Grade 3 Redness | 0 | 0 | 0 | 0
  Any Swelling | 7 | 6 | 12 | 5
  Grade 3 Swelling | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms (symp.) were headache, fever [defined as oral temperature (temp.) equal to or above 37.5 degrees Celsius (°C)], fatigue, gastrointestinal (Gastro.) symptoms [nausea, vomiting, diarrhoea and/or abdominal pain]. Any = occurrence of the symptom regardless of intensity grade and relationship. Grade 3 (G3) symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 124 | 119 | 124 | 124
Participants
  Any Fatigue | 53 | 50 | 56 | 45
  G3 Fatigue | 8 | 1 | 4 | 2
  Related Fatigue | 44 | 41 | 50 | 39
  Any Gastro. symp. | 16 | 19 | 23 | 20
  G3 Gastro. symp. | 1 | 2 | 1 | 0
  Related Gastro. symp. | 9 | 14 | 21 | 17
  Any Headache | 47 | 44 | 53 | 39
  G3 Headache | 3 | 2 | 5 | 3
  Related Headache | 37 | 33 | 39 | 33
  Any Temp. | 7 | 9 | 12 | 7
  G3 Temp. | 0 | 0 | 0 | 0
  Related Temp. | 5 | 8 | 11 | 6

3. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. "Any" was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-Day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with study vaccines administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 126 | 124 | 125 | 125
Participants | 35 | 38 | 34 | 37

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From vaccination at Day 0, up to Day 30 post-vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 126 | 124 | 125 | 125
Participants | 1 | 1 | 0 | 0

5. Primary Outcome: Titres of RSV-A Neutralizing Antibodies
Description: RSV-A neutralizing antibody titres, expressed as Geometric Mean Titres (GMTs). Seropositive subjects were defined as subjects whose antibody titre was greater than or equal to (≥) the cut-off 8 serum dilution that induced 60 % inhibition in plaque forming units (ED60).
Time Frame: At Day 0 pre-vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity which consisted of all subjects from the Total Vaccinated cohort who complied with eligibility criteria, received the study vaccine according to study procedures and had immunogenicity results in the epoch.
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 117 | 117 | 118 | 118
Titres | 397.1 [330.7 to 476.7] | 326.3 [277.1 to 384.4] | 444.2 [370.4 to 532.6] | 423.7 [360.2 to 498.4]

6. Primary Outcome: Titres of RSV-A Neutralizing Antibodies
Description: as for outcome 5
Time Frame: At Day 30 post-vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 117 | 117 | 118 | 118
Titres | 1237.0 [1094.8 to 1397.6] | 1278.7 [1141.6 to 1432.2] | 1442.5 [1287.4 to 1616.2] | 387.1 [328.4 to 456.3]

7. Secondary Outcome: Titres of RSV-A Neutralizing Antibodies
Description: RSV-A neutralizing antibody titres, expressed as Geometric Mean Titres (GMTs), were defined as any titre greater than or equal to (≥) the cut-off 8 serum dilution inducing 60 % inhibition in plaque forming units (ED60).
Time Frame: At Day 60 post-vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 109 | 111 | 108 | 111
Titres | 947.2 [832.9 to 1077.1] | 882.9 [781.9 to 996.9] | 1055.7 [926.1 to 1203.4] | 358.8 [297.8 to 432.3]

8. Secondary Outcome: Titres of RSV-A Neutralizing Antibodies
Description: as for outcome 7
Time Frame: At Day 90 post-vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 112 | 111 | 110 | 111
Titres | 837.7 [738.9 to 949.7] | 774.5 [682.6 to 878.7] | 897.5 [782.8 to 1029.2] | 358.3 [291.9 to 439.9]

9. Secondary Outcome: Concentrations of Palivizumab Competing Antibodies (PCA)
Description: Palivizumab competing antibody concentrations, expressed as Geometric Mean Concentrations (GMCs). The assay cut-off was greater than or equal to 3.34 micrograms per millilitre (µg/mL).
Time Frame: At Day 0 pre-vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 110 | 107 | 105 | 110
µg/mL | 5.4 [4.7 to 6.3] | 5.2 [4.4 to 6.0] | 4.6 [4.0 to 5.4] | 5.7 [4.8 to 6.7]

10. Secondary Outcome: Concentrations of PCA
Description: PCA concentrations, expressed as Geometric Mean Concentrations (GMCs). The assay cut-off was greater than or equal to 3.34 micrograms per millilitre (µg/mL).
Time Frame: At Day 30 post-vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 115 | 116 | 116 | 109
µg/mL | 79.9 [72.1 to 88.6] | 88.6 [79.9 to 98.2] | 97.2 [89.1 to 105.9] | 6.1 [5.3 to 7.1]

11. Secondary Outcome: Concentrations of PCA
Description: PCA concentrations, expressed as Geometric Mean Concentrations (GMCs).The assay cut-off was greater than or equal to 3.34 micrograms per millilitre (µg/mL).
Time Frame: At Day 60 post-vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 109 | 111 | 108 | 111
µg/mL | 65.9 [57.8 to 75.1] | 68.4 [61.5 to 75.9] | 74.1 [66.6 to 82.3] | 5.8 [5.0 to 6.7]

12. Secondary Outcome: Concentrations of PCA
Description: as for outcome 10
Time Frame: At Day 90 post-vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 112 | 111 | 110 | 109
µg/mL | 60.4 [54.0 to 67.6] | 62.5 [56.7 to 68.9] | 66.1 [59.9 to 73.0] | 7.5 [6.6 to 8.6]

13. Secondary Outcome: Number of Subjects With SAEs
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to study end at Day 360
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
Number analyzed (Participants) | 126 | 124 | 125 | 125
Participants | 3 | 3 | 6 | 2

ADVERSE EVENTS:
Time Frame: Solicited and Unsolicited AEs: within the 30-day (Days 0-29) post-vaccination period; SAEs: from Day 0 up to study end at Day 360.
Arm/Group | GSK3003891A 30 Non-adjuvanted Group | GSK3003891A 60 Non-adjuvanted Group | GSK3003891A 60 Adjuvanted Group | Boostrix Group
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/124 | 0/125 | 0/125
Serious Adverse Events (participants affected / at risk) | 3/126 | 3/124 | 6/125 | 2/125
Other Adverse Events (participants affected / at risk) | 93/126 | 88/124 | 112/125 | 109/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3003891A 30 Non-adjuvanted Group (N=126) | GSK3003891A 60 Non-adjuvanted Group (N=124) | GSK3003891A 60 Adjuvanted Group (N=125) | Boostrix Group (N=125)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3003891A 30 Non-adjuvanted Group (N=126) | GSK3003891A 60 Non-adjuvanted Group (N=124) | GSK3003891A 60 Adjuvanted Group (N=125) | Boostrix Group (N=125)
Gastrointestinal disorder (Gastrointestinal disorders) | 16 (16) | 19 (19) | 23 (23) | 20 (20)
Fatigue (General disorders) | 53 (53) | 50 (50) | 56 (57) | 45 (46)
Pain (General disorders) | 62 (62) | 68 (69) | 104 (105) | 104 (104)
Pyrexia (General disorders) | 7 (7) | 10 (10) | 12 (12) | 8 (8)
Swelling (General disorders) | 7 (7) | 6 (6) | 12 (12) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 7 (7) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 49 (53) | 45 (47) | 56 (59) | 41 (43)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 8 (8) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.